CLINICAL TRIAL: NCT00949910
Title: An Expanded Access Program of Tarceva (Erlotinib) in Patients With Advanced Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: An Expanded Access Program of Tarceva (Erlotinib) in Participants With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO18109; 2004-000564-28 (EudraCT Number); INC-9042 (Other: INC Research Netherlands BV)
Record Dates: First submitted 2009-04-15; First posted 2009-07-31 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Erlotinib (Experimental): Erlotinib will be given as a single agent in this expanded access program (EAP) to participants with inoperable, locally advanced, recurrent, or metastatic NSCLC. Treatment will continue until unacceptable toxicity, disease progression, or withdrawal for any other reason.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be given orally as 150 milligrams (mg) once daily until unacceptable toxicity, disease progression, or withdrawal for any other reason.
  Other Names: Tarceva

SUMMARY:
This study will provide treatment with erlotinib to participants with advanced NSCLC who have received at least one course of standard chemotherapy or radiation therapy, or who are not medically suitable for either. Efficacy and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Histologically or cytologically documented inoperable, locally advanced, metastatic, or recurrent NSCLC
* Previous treatment with no more than 2 prior chemotherapy regimens

Exclusion Criteria:

* Previous systemic anti-cancer therapy with human epidermal growth factor receptor 1 (HER1)/epidermal growth factor receptor (EGFR) inhibitors
* Inability to take oral medication
* Any other malignancies within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6586 (Actual)
Dates: Start 2004-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (395):
- Tirana, Albania
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Salta
  - Santa Fe
- Australia (16):
  - Adelaide
  - Camperdown
  - Chermside
  - Frankston
  - Fremantle
  - Geelong
  - Kurralta Park
  - Malvern
  - Melbourne
  - Perth
  - St Leonards
  - Sydney
  - Tugun
  - Waratah
  - Wodonga
  - Wollongong
- Austria (13):
  - Bludesch
  - Grimmenstein
  - Innsbruck
  - Klagenfurt
  - Kufstein
  - Leoben
  - Linz
  - Natters
  - Oberpullendorf
  - Salzburg
  - Vienna
  - Wels
  - Zams
- Belgium (32):
  - Aalst
  - Antwerp
  - Arlon
  - Baudour
  - Blankenberge
  - Borgerhout
  - Boussu
  - Brasschaat
  - Brussels
  - Charleroi
  - Edegem
  - Genk
  - Ghent
  - Gilly
  - Godinne
  - Gosselies
  - Haine-Saint-Paul
  - Hasselt
  - Kortrijk
  - Libramont
  - Liège
  - Mons
  - Namur
  - Ostend
  - Ottignies
  - Oudenaarde
  - Roeselare
  - Sint-Niklaas
  - Tielt
  - Tournai
  - Turnhout
  - Wilrijk
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo
- Brazil (17):
  - Belo Horizonte
  - Brasília
  - Campinas
  - Caxias do Sul
  - Curitiba
  - Fortaleza
  - Ijuí
  - Jaú
  - João Pessoa
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santos
  - São Paulo
  - Sorocaba
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Santiago, Chile
- China (9):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Harbin
  - Nanjing
  - Shanghai
  - Tianjin
  - Wuhan
- Colombia (2):
  - Bogotá
  - Cali
- Zagreb, Croatia
- Czechia (5):
  - Brno
  - Hradec Králové
  - Olomouc
  - Pilsen
  - Prague
- Ecuador (2):
  - Guayaquil
  - Quito
- Egypt (2):
  - Cairo
  - Giza
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (9):
  - Hämeenlinna
  - Helsinki
  - Joensuu
  - Kuopio
  - Oulu
  - Pori
  - Tampere
  - Turku
  - Vaasa
- Germany (48):
  - Amberg
  - Augsburg
  - Aurich
  - Bad Berka
  - Berlin
  - Bonn
  - Celle
  - Cologne
  - Dortmund
  - Dresden
  - Essen
  - Flensburg
  - Frankfurt
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Gauting
  - Gerlingen
  - Giessen
  - Großhansdorf
  - Halle
  - Hamburg
  - Heidelberg
  - Herne
  - Homburg/Saar
  - Kassel
  - Koblenz
  - Leipzig
  - Leverkusen
  - Lostau
  - Löwenstein
  - Lübeck
  - Mainz
  - Mannheim
  - Minden
  - Mönchengladbach
  - München
  - Neuruppin
  - Nuremberg
  - Oldenburg
  - Osnabrück
  - Rostock
  - Saarbrücken
  - Trier
  - Ulm
  - Wangen
  - Wiesbaden
  - Wuppertal
  - Würselen
- Greece (5):
  - Athens
  - Haidari
  - Heraklion
  - Neo Faliro
  - Thessaloniki
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Hungary (7):
  - Budapest
  - Deszk
  - Kecskemét
  - Mátraháza
  - Nyíregyháza
  - Pécs
  - Törökbálint
- India (4):
  - Bangalore
  - New Delhi
  - Pune
  - Vellore
- Jakarta, Indonesia
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Israel (13):
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Safed
  - Tel Aviv
  - Ẕerifin
- Italy (46):
  - Ancona
  - Avellino
  - Aviano
  - Bari
  - Benevento
  - Bergamo
  - Bollate
  - Bologna
  - Brescia
  - Candiolo
  - Catania
  - Catanzaro
  - Cosenza
  - Cuneo
  - Fabriano
  - Feltre - Bl
  - Florence
  - Genova
  - La Spezia
  - Lido di Camaiore
  - Livorno
  - Meldola
  - Messina
  - Milan
  - Mirano
  - Modena
  - Napoli
  - Nuoro
  - Orbassano
  - Palermo
  - Parma
  - Pavia
  - Perugia
  - Pescara
  - Pisa
  - Rionero in Vulture
  - Roma
  - Salerno
  - San Giovanni Rotondo
  - Sassari
  - Siena
  - Sondrio
  - Taormina
  - Torino
  - Trento
  - Udine
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Kuala Lumpur, Malaysia
- Mexico (18):
  - Acapulco
  - Chihuahua City
  - Guadalajara
  - Juárez
  - León
  - Matamoros
  - Mexicali
  - Mexico City
  - Mérida
  - Monterrey
  - Obregón
  - Puebla City
  - San Luis Potosí City
  - Tampico
  - Tijuana
  - Toluca
  - Torreón
  - Zapopan
- Netherlands (36):
  - 's-Hertogenbosch
  - Alkmaar
  - Amersfoort
  - Amstelveen
  - Amsterdam
  - Arnhem
  - Assen
  - Beverwijk
  - Boxmeer
  - Breda
  - Capelle Ad Yssel
  - Drachten
  - Eindhoven
  - Enschede
  - Flushing
  - Groningen
  - Haarlem
  - Harderwijk
  - Heerlen
  - Helmond
  - Hengelo
  - Hoofddorp
  - Leiden
  - Leiderdorp
  - Maastricht
  - Nieuwegein
  - Nijmegen
  - Roermond
  - Rotterdam
  - Sliedrecht
  - The Hague
  - Veldhoven
  - Venlo
  - Vlaardingen
  - Zaandam
  - Zwolle
- New Zealand (4):
  - Christchurch
  - Hamilton
  - Palmerston North
  - Wellington
- Panama City, Panama
- Peru (2):
  - Callao
  - Lima
- Poland (7):
  - Gdansk
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
  - Wroclaw
  - Zabrze
- Portugal (5):
  - Lisbon
  - Porto
  - São Martinho do Bispo
  - Setúbal
  - Vila Nova de Gaia
- Romania (8):
  - Alba Iulia
  - Baia Mare
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Sibiu
  - Suceava
  - Timișoara
- Russia (12):
  - Barnaul
  - Kazan'
  - Krasnodar
  - Moscow
  - Obninsk
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
  - Tyumen
  - Ufa
  - Volgograd
- Riyadh, Saudi Arabia
- Serbia (2):
  - Belgrade
  - Novi Sad
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Nitra
  - Poprad
- Ljubljana, Slovenia
- South Korea (12):
  - Bundang City
  - Busan
  - Cheonan
  - Daegu
  - Daejeon
  - Gwangju
  - Iksan
  - Incheon
  - Kyunggi-do
  - Pusan
  - Seoul
  - Suwon
- Sweden (7):
  - Falun
  - Gothenburg
  - Linköping
  - Lund
  - Malmo
  - Stockholm
  - Uppsala
- Switzerland (6):
  - Aarau
  - Baden
  - Chur
  - Locarno
  - Lucerne
  - Zurich
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Shhiye, Ankara
- Montevideo, Uruguay
- Caracas, Venezuela

REFERENCES:
- [Derived] Huang Y, Zhang L, Shi Y, Ma S, Liao M, Bai C, Zhang Q, Wang C, Luo F, Yu S, Qin S, Zhi X, Zhou C. Efficacy of erlotinib in previously treated patients with advanced non-small cell lung cancer: analysis of the Chinese subpopulation in the TRUST study. Jpn J Clin Oncol. 2015 Jun;45(6):569-75. doi: 10.1093/jjco/hyv036. Epub 2015 Apr 7. PMID 25855621
- [Derived] Heigener DF, Wu YL, van Zandwijk N, Mali P, Horwood K, Reck M. Second-line erlotinib in patients with advanced non-small-cell lung cancer: subgroup analyses from the TRUST study. Lung Cancer. 2011 Nov;74(2):274-9. doi: 10.1016/j.lungcan.2011.02.017. Epub 2011 Mar 24. PMID 21439671

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Erlotinib was given as a single agent in this expanded access program (EAP) to participants with inoperable, locally advanced, recurrent, or metastatic non-small cell lung cancer (NSCLC). Participants were treated with 150 milligrams (mg) oral erlotinib once daily until unacceptable toxicity, disease progression, or withdrawal for any other reason. The dose could be reduced in the event of toxicity, and some participants therefore received 50 or 100 mg once daily. The study completed after every participant had either died or been followed for 6 months after stopping erlotinib.
Period: Overall Study
Arm/Group | Erlotinib
Started | 6586
Completed | 10
Not Completed | 6576
Not completed — Progressive Disease | 3750
Not completed — Symptomatic Deterioration | 1088
Not completed — Lost to Follow-up | 100
Not completed — Study Drug-Related Adverse Event | 315
Not completed — Participant Refusal | 390
Not completed — Death Due to Malignant Disease | 456
Not completed — Death Due to Progression/Deterioration | 4
Not completed — Death Due to Adverse Event | 115
Not completed — Death Due to Toxicity | 3
Not completed — Death from Unknown Cause | 5
Not completed — Unspecified Progression/Deterioration | 13
Not completed — Switched to Compassionate/Other Use | 174
Not completed — Switched to Commercial Treatment | 4
Not completed — Violation of Eligibility | 23
Not completed — Logistical Reasons | 13
Not completed — Non-Compliance | 10
Not completed — Prolonged Dosing Interruption | 4
Not completed — Adverse Event | 83
Not completed — Serious Adverse Event | 6
Not completed — Physician/Participant Decision | 7
Not completed — Other | 4
Not completed — No Data | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT)/Safety Population: All participants who received at least one dose of erlotinib.
Groups:
- Erlotinib: Erlotinib was given as a single agent in this EAP to participants with inoperable, locally advanced, recurrent, or metastatic NSCLC. Participants were treated with 150 mg oral erlotinib once daily until unacceptable toxicity, disease progression, or withdrawal for any other reason. The dose could be reduced in the event of toxicity, and some participants therefore received 50 or 100 mg once daily. The study completed after every participant had either died or been followed for 6 months after stopping erlotinib.
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2608
  Male | 3978

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response was defined as a best overall response of either complete response (CR) or partial response (PR) as assessed by RECIST during the study. CR was defined as disappearance of all clinical and radiographic evidence of target and non-target lesions, normal tumor markers, and absence of tumor-related symptoms. PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥28 days after the initial assessment of CR or PR. The percentage of participants (in nearest integer) with objective response was reported.
Time Frame: Up to approximately 4.5 years; assessed at Baseline, according to institutional standards during treatment (up to 3.5 years), and every 6 months thereafter
Population: ITT/Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
percentage of participants | 11

2. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST
Description: Disease control was defined as a best overall response of either CR, PR, or stable disease (SD) as assessed by RECIST during the study. CR was defined as disappearance of all clinical and radiographic evidence of target and non-target lesions, normal tumor markers, and absence of tumor-related symptoms. PR was defined as ≥30% decrease in sum LD of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥28 days after the initial assessment of CR or PR. SD was defined as neither sufficient shrinkage to qualify for PR but less than (<) 20% increase in sum LD. The percentage of participants (in nearest integer) with disease control was reported.
Time Frame: as for outcome 1
Population: ITT/Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
percentage of participants | 56

3. Secondary Outcome: Percentage of Participants by Best Overall Response According to RECIST
Description: Tumor response was assessed by RECIST during the study. CR was defined as disappearance of all clinical and radiographic evidence of target and non-target lesions, normal tumor markers, and absence of tumor-related symptoms. PR was defined as ≥30% decrease in sum LD of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥28 days after the initial assessment of CR or PR. SD was defined as neither sufficient shrinkage to qualify for PR but <20% increase in sum LD. Disease progression or progressive disease (PD) was defined as ≥20% increase in sum LD in reference to the smallest on-treatment sum LD, or the appearance of new lesions. The percentage of participants (in nearest integer unless the percentage is <1) with each type of best overall response was reported.
Time Frame: as for outcome 1
Population: ITT/Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
percentage of participants
  Complete Response (CR) | 0.7
  Partial Response (PR) | 10
  Stable Disease (SD) | 45
  Progressive Disease (PD) | 23
  Not Evaluable | 3
  Not Done | 18
  Not Known | 0.0
  No Data | 0.3

4. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to RECIST
Description: Tumor response was assessed by RECIST during the study. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-treatment sum LD, or the appearance of new lesions. The percentage of participants (in nearest integer) who died or experienced PD was reported.
Time Frame: as for outcome 1
Population: ITT/Safety Population; only participants with available data were included.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6580
percentage of participants | 93

5. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST
Description: Tumor response was assessed by RECIST during the study. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-treatment sum LD, or the appearance of new lesions. PFS was defined as the time from start of treatment to the first event of death or PD. The median duration of PFS and corresponding 95% confidence interval (CI) were estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: as for outcome 1
Population: ITT/Safety Population; only participants with available data were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 6580
months | 3.3 [3.1 to 3.4]

6. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants (in nearest integer) who died from any cause was reported.
Time Frame: Up to approximately 4.5 years; assessed continuously during treatment (up to 3.5 years) and every 6 months thereafter
Population: ITT/Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
percentage of participants | 81

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of treatment to date of death for any reason. The median duration of OS and corresponding 95% CI were estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: Up to approximately 4.5 years; assessed continuously during treatment (up to 3.5 years) and every 6 months thereafter
Population: ITT/Safety Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 6586
months | 7.9 [7.6 to 8.3]

ADVERSE EVENTS:
Time Frame: Up to approximately 4.5 years; assessed continuously during treatment (up to 3.5 years) and every 6 months thereafter
Description: ITT/Safety Population. As planned only unexpected erlotinib-related adverse events (AEs) and erlotinib-related rash were to be reported, with the exception of serious adverse events (SAEs) and AEs leading to premature withdrawal which were collected regardless of causality.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 2983/6586
Other Adverse Events (participants affected / at risk) | 0/6586
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=6586)
Anaemia (Blood and lymphatic system disorders) | 43
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 12
Angina pectoris (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 13
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 12
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 9
Cardio-respiratory distress (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 14
Cor pulmonale (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Hypertensive heart disease (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 18
Myocardial ischaemia (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 20
Pericarditis (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 3
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 5
Conjunctivitis (Eye disorders) | 2
Diplopia (Eye disorders) | 2
Iridocele (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Visual disturbance (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 32
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 6
Acute abdomen (Gastrointestinal disorders) | 3
Appendicitis perforated (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 6
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 83
Diverticular perforation (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 21
Enteritis (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2
Gastric perforation (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Gastritis erosive (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 19
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gastrointestinal ulcer perforation (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 6
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 8
Inguinal hernia (Gastrointestinal disorders) | 3
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 5
Intestinal perforation (Gastrointestinal disorders) | 2
Jejunal perforation (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 35
Necrotising oesophagitis (Gastrointestinal disorders) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal spasm (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 3
Rectal polyp (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 5
Subileus (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 45
Asthenia (General disorders) | 18
Catheter related complication (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 51
Condition aggravated (General disorders) | 2
Death (General disorders) | 14
Disease progression (General disorders) | 292
Drug withdrawal syndrome (General disorders) | 1
Euthanasia (General disorders) | 2
Fatigue (General disorders) | 16
Gait disturbance (General disorders) | 3
General physical health deterioration (General disorders) | 195
Hyperpyrexia (General disorders) | 1
Ill-defined disorder (General disorders) | 14
Local swelling (General disorders) | 1
Malaise (General disorders) | 7
Mucosal inflammation (General disorders) | 3
Multi-organ failure (General disorders) | 3
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 33
Performance status decreased (General disorders) | 8
Pyrexia (General disorders) | 52
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 2
Ulcer (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 4
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hepatic pain (Hepatobiliary disorders) | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 5
Liver disorder (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 14
Bronchitis bacterial (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 12
Bursitis infective (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Catheter sepsis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Central line infection (Infections and infestations) | 6
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Diabetic gangrene (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Empyema (Infections and infestations) | 4
Enterocolitis infectious (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 3
Extradural abscess (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 15
Gastrointestinal infection (Infections and infestations) | 2
Groin abscess (Infections and infestations) | 1
Herpangina (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infected epidermal cyst (Infections and infestations) | 1
Infection (Infections and infestations) | 23
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 20
Lung abscess (Infections and infestations) | 2
Lung infection (Infections and infestations) | 12
Lung infection pseudomonal (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 217
Pneumonia primary atypical (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 14
Sepsis (Infections and infestations) | 17
Septic shock (Infections and infestations) | 6
Sinobronchitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 12
Urosepsis (Infections and infestations) | 2
Vulval abscess (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 7
Femur fracture (Injury, poisoning and procedural complications) | 6
Fracture (Injury, poisoning and procedural complications) | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 3
Hip fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 8
Joint dislocation (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Wound complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Aspiration pleural cavity (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Bronchoalveolar lavage (Investigations) | 1
Drug level increased (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 2
International normalised ratio abnormal (Investigations) | 1
International normalised ratio increased (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Pulmonary function test decreased (Investigations) | 1
Sigmoidoscopy (Investigations) | 1
Weight decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 12
Cachexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 29
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Malnutrition (Metabolism and nutrition disorders) | 1
Oral intake reduced (Metabolism and nutrition disorders) | 2
Tetany (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 36
Bone pain (Musculoskeletal and connective tissue disorders) | 26
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Dactylitis (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Pathological fracture (Musculoskeletal and connective tissue disorders) | 7
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 54
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 810
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Non-small cell lung cancer Stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Altered state of consciousness (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 5
Ataxia (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 5
Cerebral haemorrhage (Nervous system disorders) | 4
Cerebral infarction (Nervous system disorders) | 11
Cerebral ischaemia (Nervous system disorders) | 4
Cerebrovascular accident (Nervous system disorders) | 24
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 13
Depressed level of consciousness (Nervous system disorders) | 2
Diplegia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 4
Facial paresis (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hemiparesis (Nervous system disorders) | 6
Hemiplegia (Nervous system disorders) | 4
Hepatic encephalopathy (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Meningeal disorder (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 3
Monoplegia (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Paraparesis (Nervous system disorders) | 4
Paraplegia (Nervous system disorders) | 3
Partial seizures (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral paralysis (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Psychomotor skills impaired (Nervous system disorders) | 1
Quadriplegia (Nervous system disorders) | 1
Radicular pain (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 12
Spinal cord disorder (Nervous system disorders) | 1
Subdural hygroma (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 19
Syncope vasovagal (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 7
Agitation (Psychiatric disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 26
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 6
Disorientation (Psychiatric disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Vomiting psychogenic (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Glomerulosclerosis (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 7
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 6
Renal failure acute (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 5
Cervical polyp (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 340
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 83
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 107
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleurocutaneous fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 68
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 115
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 32
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1
Angioplasty (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Jaw operation (Surgical and medical procedures) | 1
Pain management (Surgical and medical procedures) | 1
Pleurodesis (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Renal stone removal (Surgical and medical procedures) | 1
Spinal decompression (Surgical and medical procedures) | 1
Thoracic cavity drainage (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 2
Aortic aneurysm rupture (Vascular disorders) | 1
Arterial insufficiency (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Arterial thrombosis (Vascular disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 4
Axillary vein thrombosis (Vascular disorders) | 2
Cardiovascular insufficiency (Vascular disorders) | 3
Circulatory collapse (Vascular disorders) | 5
Deep vein thrombosis (Vascular disorders) | 31
Embolism (Vascular disorders) | 4
Haemorrhage (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 2
Ischaemia (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Macroangiopathy (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2
Pelvic venous thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 2
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Subclavian artery stenosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 2
Superior vena caval occlusion (Vascular disorders) | 11
Thrombophlebitis (Vascular disorders) | 2
Thrombophlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 7
Vascular rupture (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Venous occlusion (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.